CLINICAL TRIAL: NCT06142097
Title: Sensor Technology Assessments of Reproductive Target Study
Acronym: START
Status: Completed | Type: Observational
Sponsor: Ouraring Inc. (Industry)
Collaborators: UCSF Center for Reproductive Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: OS22WH01
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Menstrual Cycle; Ovulation; Menstruation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study was to better understand female reproductive health in the context of using wearable technology. Participants were provided and wore an Oura Ring, tracked their menstrual cycles, provided at-home ovulation test results, and had their cycles monitored via trans-vaginal ultrasounds. The study aimed to collect data from females with regular menstrual cycles.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women age 18-42 years
* Regular menstrual cycles every 25-32 days
* Own an iPhone or Android mobile device
* Agree to follow study protocol such as wearing the Oura Ring for the duration of the study, at-home ovulation testing, present for frequent ultrasounds

Exclusion Criteria:

* Non-English speaking
* Current use of hormonally active medications
* History of infertility
* History of recurrent pregnancy loss
* Current circadian disruptions

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Convenience sampling of individuals willing to travel to clinic and who meet other criteria
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Retrospective ovulation day | 6 months
Prospective ovulation day | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Jaswa, M.D., M.Sc., Principal Investigator — UCSF Center for Reproductive Health
Locations (1):
- UCSF Center for Reproductive Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No